CLINICAL TRIAL: NCT01483326
Title: FAct: A Non-interventional Multi-center Study to Follow Patients Starting With RoActemra Assessing the Long Term Efficacy, Effectiveness and Safety of RoActemra
Brief Title: An Observational Study on Long-Term Efficacy and Safety of RoActemra/Actemra (Tocilizumab) in Patients With Moderate to Severe Rheumatoid Arthritis (FAct)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25411
Record Dates: First submitted 2011-11-23; First posted 2011-12-01 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the long-term efficacy and safety of RoActemra/Actemra (tocilizumab in participants of the ACT SURE clinical trial and further patients with moderate to severe rheumatoid arthritis starting or receiving RoActemra/Actemra. Data will be collected from each patient for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >18 years of age
* Participants in the ACT-SURE trial, or patients with moderate to severe rheumatoid arthritis starting or receiving RoActemra/Actemra

Exclusion Criteria:

* Contra-indications for RoActemra/Actemra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the ACT SURE clinical trial or patients with moderate to severe rheumatoid arthritis starting or receiving RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2010-12-31 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Change in disease activity score (DAS 28) | baseline and up to 4 years

SECONDARY OUTCOMES:
Change in disability, assessed by Health Assessment Questionnaire (HAQ) | baseline and up to 4 years
Change in concomitant medication (especially tapering of steroids) | baseline and up to 4 years
Change in dosage schedule (modification/interruption/discontinuation) | baseline and up to 4 years
Safety: Incidence of adverse events | up to 4 years
Response (DAS 28) according to patient-related factors (C-reactive protein, rheumatoid factor, inadequate response to anti-TNF/DMARDs, duration of illness) | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Netherlands (19):
  - Jan Van Breemen Instituut, Amsterdam
  - Gelre Ziekenhuis; Reumatology, Apeldoorn
  - Rijnstate Ziekenhuis; Afdeling Reumatologie, Arnhem
  - Amphia ziekenhuis, locatie langendijk, Breda
  - Deventer ziekenhuis, Deventer
  - MC groep - locatie Emmeloord, Emmeloord
  - Scheper Ziekenhuis, Emmen
  - Medisch Centrum Twente; Rheumatology, Enschede
  - Ziekenhuis Walcheren; Reumatologie, Flushing
  - Groene Hart Ziekenhuis, Gouda
  - Röpcke Zweers ziekenhuis; Reumatologie, Hardenberg
  - Tergooiziekenhuizen, loc. Hilversum, Hilversum
  - Medisch Centrum Leeuwarden; Reumatology, Leeuwarden
  - Maastricht University Medical Centre; Rheumatology, Maastricht
  - St. Antonius Ziekenhuis; Pharmacy, Nieuwegein
  - St. Maartenskliniek, Nijmegen
  - Maasstadziekenhuis; Reumatologie, Rotterdam
  - Vlietland Hospital, Schiedam
  - Leyenburg Ziekenhuis; Internal Medecine, The Hague